CLINICAL TRIAL: NCT01749540
Title: A Phase 2, Open-Label, Ascending Dose Study to Evaluate the Effects of ACE-536 in Patients With β-Thalassemia
Brief Title: Study to Evaluate the Safety and Efficacy of Luspatercept (ACE-536) in Participants With Beta-thalassemia (A536-04/MK-6143-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A536-04; MK-6143-002 (Other: Merck); A536-04 (Other: Acceleron); 2012-002499-15 (EudraCT Number)
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: B-Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Luspatercept 0.2 mg/kg (Experimental): Participants receive luspatercept 0.2 mg/kg as a subcutaneous (SC) injection every 3 weeks (Q3W) on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: luspatercept
- Luspatercept 0.4 mg/kg (Experimental): Participants receive luspatercept 0.4 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: luspatercept
- Luspatercept 0.6 mg/kg (Experimental): Participants receive luspatercept 0.6 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: luspatercept
- Luspatercept 0.8 mg/kg (Experimental): Participants receive luspatercept 0.8 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: luspatercept
- Luspatercept 1.0 mg/kg (Experimental): Participants receive luspatercept 1.0 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: luspatercept
- Luspatercept 1.25 mg/kg (Experimental): Participants receive luspatercept 1.25 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
  Interventions: Drug: luspatercept
- Expansion Cohort (Experimental): Participants receive an initial dose of luspatercept 0.8 mg/kg as an SC injection on Day 1 of Cycle 1 (Cycle length = 21 days). For each subsequent cycle (up to 5 cycles), the dose was titrated up to a maximum dose of 1.25 mg/kg based on the safety review team (SRT) recommendations.
  Interventions: Drug: luspatercept

INTERVENTIONS:
Drug: luspatercept — subcutaneous injection
  Other Names: ACE-536; MK-6143

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics, of ascending doses of luspatercept in participants with β-thalassemia.

The primary objective of this study is to evaluate erythroid response, defined as:

1. a hemoglobin increase of ≥ 1.5 g/dL from baseline for ≥ 14 days (in the absence of red blood cell [RBC] transfusions) in non-transfusion dependent participants, or
2. a ≥ 20% reduction in RBC transfusion burden compared to pretreatment in transfusion dependent participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Men or women ≥18 years of age
* For the dose escalation phase of the study: documented diagnosis of β-thalassemia intermedia (transfusion dependent participants must not have begun regular transfusions at age <4.0 years). For the expansion cohort: documented diagnosis of β-thalassemia (including β-thalassemia major or β-thalassemia intermedia)
* Prior splenectomy or spleen size <18 cm in the longest diameter by abdominal ultrasound (dose escalation cohorts only)
* Anemia, defined as: (1) mean hemoglobin concentration <10.0 g/dL of 2 measurements (one performed within one day prior to Cycle 1 Day 1 and the other performed during the screening period [Day -28 to Day -1]) in non-transfusion dependent participants, defined as having received < 4 units of RBCs within 8 weeks prior to Cycle 1 Day 1, or (2) transfusion dependent participants, defined as requiring ≥ 4 units of RBCs every 8 weeks (confirmed over 6 months prior to Cycle 1 Day 1)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <3 x upper limit of normal (ULN)
* Serum creatinine ≤1.5 x ULN
* Adequate pregnancy avoidance measures
* Participants are able to adhere to the study visit schedule, understand, and comply with all protocol requirements
* Understand and able to provide written informed consent

Key Exclusion Criteria:

* Any clinically significant pulmonary (including pulmonary hypertension), cardiovascular, endocrine, neurologic, hepatic, gastrointestinal, infectious, immunological (including clinically significant allo- or auto-immunization) or genitourinary disease considered by the investigator as not adequately controlled prior to Cycle 1 Day 1
* Folate deficiency
* Symptomatic splenomegaly
* Known positive for human immunodeficiency virus (HIV), active infectious hepatitis B virus (HBV) or active infectious hepatitis C virus (HCV)
* Known history of thromboembolic events ≥Grade 3 according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 (current active minor version)
* Ejection fraction <50% by echocardiogram, multi-gated acquisition scan (MUGA), or cardiac magnetic resonance imaging (MRI)
* Uncontrolled hypertension defined as systolic blood pressure (BP) ≥150 mm Hg or diastolic BP ≥95 mm Hg
* Heart failure class 3 or higher (New York Heart Association [NYHA])
* QTc >450 msec on screening electrocardiogram (ECG)
* Platelet count <100 x10^9/L or >1,000 x10^9/L
* Proteinuria ≥Grade 2
* Any active infection requiring parenteral antibiotic therapy within 28 days prior to Cycle 1 Day 1 or oral antibiotics within 14 days of Cycle 1 Day 1
* Treatment with another investigational drug or device, or approved therapy for investigational use ≤28 days prior to Cycle 1 Day 1, or if the half-life of the previous investigational product is known, within 5 times the half-life prior to Cycle 1 Day 1, whichever is longer
* Transfusion event within 7 days prior to Cycle 1 Day 1
* Participants receiving or planning to receive hydroxyurea treatment. Participants must not have had hydroxyurea within 90 days of Cycle 1 Day 1
* Splenectomy within 56 days prior to Cycle 1 Day 1
* Major surgery (except splenectomy) within 28 days prior to Cycle 1 Day 1. Participants must have completely recovered from any previous surgery prior to Cycle 1 Day 1
* Iron chelation therapy initiated within 56 days prior to Cycle 1 Day 1
* Cytotoxic agents, systemic corticosteroids, immunosuppressants, or anticoagulant therapy such as warfarin or heparin within 28 days prior to Cycle 1 Day 1 (prophylactic aspirin up to 100 mg/day is permitted)
* Pregnant or lactating women
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational drug
* Prior treatment with sotatercept (ACE-011) or luspatercept (ACE-536)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-02-28 (Actual); Primary Completion 2015-11-11 (Actual); Study Completion 2015-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- Laiko General Hospital, Ampelokipi, Athens, Greece
- Italy (7):
  - Ospedale "A. Perriino" U.O Ematologia, Brindisi
  - ARNAS Garibaldi - P.O. Garibaldi Centro, Catania
  - A.O.U. Arcispedale S. Anna, Ferrara
  - CEMEF Medicina 2, Modena
  - A.O.U. Seconda Università degli Studi di Napoli, Napoli
  - AORN A. Cardarelli, Napoli
  - A.O.U. San Luigi Gonzaga, Orbassano

REFERENCES:
- [Derived] Piga A, Longo F, Gamberini MR, Voskaridou E, Ricchi P, Caruso V, Pietrangelo A, Zhang X, Shetty JK, Attie KM, Tartaglione I. Long-term safety and erythroid response with luspatercept treatment in patients with beta-thalassemia. Ther Adv Hematol. 2022 Dec 5;13:20406207221134404. doi: 10.1177/20406207221134404. eCollection 2022. PMID 36505885
- [Derived] Cappellini MD, Taher AT. The use of luspatercept for thalassemia in adults. Blood Adv. 2021 Jan 12;5(1):326-333. doi: 10.1182/bloodadvances.2020002725. PMID 33570654
- [Derived] Piga A, Perrotta S, Gamberini MR, Voskaridou E, Melpignano A, Filosa A, Caruso V, Pietrangelo A, Longo F, Tartaglione I, Borgna-Pignatti C, Zhang X, Laadem A, Sherman ML, Attie KM. Luspatercept improves hemoglobin levels and blood transfusion requirements in a study of patients with beta-thalassemia. Blood. 2019 Mar 21;133(12):1279-1289. doi: 10.1182/blood-2018-10-879247. Epub 2019 Jan 7. PMID 30617198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from the study A536-04 were eligible to be initiated in extension study A536-06 (NCT02268409) following the last dose of luspatercept. Participants did not undergo an end of study visit in study A536-04 but instead were initiated immediately into the extension study.
Groups:
- Luspatercept 0.2 mg/kg: Participants received luspatercept 0.2 mg/kg as a subcutaneous (SC) injection every 3 weeks (Q3W) on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.4 mg/kg: Participants received luspatercept 0.4 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.6 mg/kg: Participants received luspatercept 0.6 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 0.8 mg/kg: Participants received luspatercept 0.8 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.0 mg/kg: Participants received luspatercept 1.0 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept 1.25 mg/kg: Participants received luspatercept 1.25 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Expansion Cohort: Participants received an initial dose of luspatercept 0.8 mg/kg as an SC injection on Day 1 of Cycle 1 (Cycle length = 21 days). For each subsequent cycle (up to 5 cycles), the dose was titrated up to a maximum dose of 1.25 mg/kg based on the safety review team (SRT) recommendations.
Period: Overall Study
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Started | 6 | 6 | 6 | 6 | 6 | 5 | 29
Completed | 6 | 6 | 6 | 5 | 6 | 2 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 3 | 25
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Initiated into extension study A536-06 | 0 | 0 | 0 | 0 | 0 | 2 | 24

BASELINE CHARACTERISTICS:
Population: All randomized participants who received ≥1 dose of study treatment
Groups:
- Luspatercept 0.2 mg/kg: Participants received luspatercept 0.2 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Total: Total of all reporting groups
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.3 (11.3) | 32.0 (7.1) | 39.2 (12.4) | 33.2 (10.3) | 40.8 (11.9) | 42.8 (7.9) | 38.9 (10.9) | 38.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 5 | 2 | 4 | 13 | 31
  Male | 2 | 5 | 4 | 1 | 4 | 1 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 5 | 29 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 6 | 6 | 6 | 5 | 6 | 5 | 28 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline for ≥14 Days
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline for ≥14 days in the absence of blood transfusion. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period. Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion or 56 days after the last dose were excluded from analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline for ≥14 days is presented.
Time Frame: Up to approximately 20 weeks
Population: All participants who received ≥1 dose of study treatment and received <4 units of RBCs within 8 weeks prior to the first dose of study drug and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 3 | 2 | 1 | 10
Percentage of participants | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 52.2] | 66.7 [9.4 to 99.2] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 60.0 [26.2 to 87.8]

2. Primary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥20% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 12-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). The interval during the pretreatment period was defined as the 12 weeks prior to the first dose of study drug. An interval during the treatment plus follow-up period was defined as any 12-week interval after the first dose of study drug. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥20% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 weeks)
Population: All participants who received ≥1 dose of study treatment and received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug) and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 4 | 19
Percentage of participants |  |  | 100 [2.5 to 100] | 66.7 [9.4 to 99.2] | 100 [39.8 to 100] | 75.0 [19.4 to 99.4] | 78.9 [54.4 to 93.9]

3. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 20 weeks
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
Participants | 5 | 6 | 5 | 6 | 6 | 5 | 26

4. Secondary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Description: An SAE was any adverse event, occurring at any dose level/regimen and regardless of causality that: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect; or was an important medical event. The number of participants who experienced an SAE is presented.
Time Frame: Up to approximately 20 weeks
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE) of Grade 3 or Greater
Description: AEs were graded using the National Cancer Institute Common Toxicity Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0) and graded as follows: Grade 1=mild; Grade 2=moderate; Grade 3=severe or medically significant but not immediately life-threatening; Grade 4=life-threatening consequences; and Grade 5=death related to AE. An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who experienced an AE of ≥Grade 3 is presented.
Time Frame: Up to approximately 20 weeks
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
Participants | 0 | 1 | 0 | 1 | 2 | 0 | 4

6. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due To an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it is considered related to the study drug. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 12 weeks
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
Participants | 0 | 0 | 1 | 2 | 0 | 0 | 2

7. Secondary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: DLTs were determined using the National Cancer Institute Common Toxicity Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0) and graded as follows: Grade 1=mild; Grade 2=moderate; Grade 3=severe or medically significant but not immediately life-threatening; Grade 4=life-threatening consequences; and Grade 5=death related to AE. The occurrence of any of the following toxicities occurring up to 28 days after the first dose was considered a DLT: treatment-related serious adverse event (SAE) ≥ Grade 3; treatment related non-hematologic adverse event (AE) ≥ Grade 3; and treatment related hematologic AE ≥ Grade 4. The number of participants who experienced a DLT is presented.
Time Frame: Up to 28 days
Population: The DLT analysis population consisted of all participants who received ≥1 dose of study treatment and were observed for DLTs for 28 days after the first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.0 g/dL From Baseline During a Rolling 8-week Interval
Description: A modified erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.0 g/dL from baseline during an 8-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period. Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion or 56 days after the last dose were excluded from analysis. NTD participants were participants who had received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug. An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.0 g/dL from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 20 Weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 3 | 2 | 1 | 10
Percentage of participants | 16.7 [0.4 to 64.1] | 16.7 [0.4 to 64.1] | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 70.0 [34.8 to 93.3]

9. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline During a Rolling 8-week Interval
Description: A modified erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline during an 8-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period. Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion or 56 days after the last dose were excluded from analysis. NTD participants were participants who had received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug. An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 20 Weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 3 | 2 | 1 | 10
Percentage of participants | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 52.2] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 60.0 [26.2 to 87.8]

10. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.0 g/dL From Baseline During a Rolling 12-week Interval
Description: A modified erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.0 g/dL from baseline during a 12-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period. Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion or 56 days after the last dose were excluded from analysis. NTD participants were participants who had received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug. A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.0 g/dL from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 Weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 3 | 2 | 1 | 10
Percentage of participants | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 45.9] | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 60.0 [26.2 to 87.8]

11. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline During a Rolling 12-week Interval
Description: A modified erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline during a 12-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period. Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion or 56 days after the last dose were excluded from analysis. NTD participants were participants who had received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug. A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 Weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 3 | 2 | 1 | 10
Percentage of participants | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 52.2] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 50.0 [18.7 to 81.3]

12. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥50% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 8-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during an 8-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a ≥50% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 20 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 4 | 19
Percentage of participants |  |  | 100 [2.5 to 100] | 100 [29.2 to 100] | 100 [39.8 to 100] | 75.0 [19.4 to 99.4] | 78.9 [54.4 to 93.9]

13. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥50% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 12-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a ≥50% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 4 | 19
Percentage of participants |  |  | 100 [2.5 to 100] | 66.7 [9.4 to 99.2] | 100 [39.8 to 100] | 50.0 [6.8 to 93.2] | 42.1 [20.3 to 66.5]

14. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants Who Maintained Red Blood Cell (RBC) Transfusion Independence For ≥8 Weeks
Description: Transfusion independence for TD participants was defined as the percentage of participants who did not require RBC transfusion units (or milliliters) transfused for ≥8 weeks in the study after start of treatment. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants who maintained transfusion independence for ≥8 weeks is presented.
Time Frame: Any 8-week interval during the study (up to approximately 20 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 4 | 4 | 19
Percentage of participants |  |  | 100 [2.5 to 100] | 0.0 [0.0 to 70.8] | 75.0 [19.4 to 99.4] | 0.0 [0.0 to 60.2] | 10.5 [1.3 to 33.1]

15. Secondary Outcome: Time To Erythroid Response for Non-transfusion Dependent (NTD) Participants Who Achieved a Hemoglobin Increase ≥1.0 g/dL During a Rolling 12-week Interval by Pooled Dose Groups
Description: Time to erythroid response was defined as the time from first dose to the first date of any rolling 12-week window achieving a hemoglobin increase ≥1.0 g/dL. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by analysis cutoff were censored. The time to the first date of any rolling 12-week window achieving a hemoglobin increase ≥1.0 g/dL is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 weeks)
Population: All participants who received ≥1 dose of study treatment and received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug and had data available for the analyses. As defined in the clinical study report, the participants with response were pooled into low and high dose groups to reduce the variation of the analyses.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Luspatercept Low Dose Group: 0.2 to 0.4 mg/kg: Participants received luspatercept 0.2 or 0.4 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
- Luspatercept High Dose Group: 0.6 to 1.25 mg/kg: Participants received luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg as an SC injection Q3W on Day 1 of each cycle for up to 5 cycles (each cycle length = 21 days).
Arm/Group | Luspatercept Low Dose Group: 0.2 to 0.4 mg/kg | Luspatercept High Dose Group: 0.6 to 1.25 mg/kg
Number analyzed (Participants) | 1 | 13
Days | 8.0 (NA) — NA=standard deviation cannot be calculated for 1 participant. | 9.9 (6.29)

16. Secondary Outcome: Time To Erythroid Response for Transfusion Dependent (TD) Participants Who Achieved a Transfusion Burden Reduction of ≥50% During a Rolling 12-week Interval
Description: Time to erythroid response was defined as the time from the first dose to the first date of any rolling 12-week window achieving a red blood cell (RBC) transfusion burden reduction of ≥50% compared to pretreatment. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by analysis cutoff were censored. The time to the first date of any rolling 12-week window achieving a red blood cell transfusion burden reduction of ≥50% compared to pretreatment is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 weeks)
Population: All participants who received ≥1 dose of study treatment and have received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug) and had data available for the analyses. As defined in the clinical study report, the participants with response were pooled into low and high dose groups to reduce the variation of the analyses.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Low Dose Group: 0.2 to 0.4 mg/kg | Luspatercept High Dose Group: 0.6 to 1.25 mg/kg
Number analyzed (Participants) | 0 | 17
Days |  | 4.8 (8.30)

17. Secondary Outcome: Duration of Erythroid Response for Non-transfusion Dependent (NTD) Participants Who Achieved a Hemoglobin Increase ≥1.0 g/dL During a Rolling 12-week Interval
Description: Duration of erythroid response was defined as the time from the first rolling 12-week window achieving a hemoglobin increase of ≥1.0 g/dL to the date of the last consecutive rolling 12-week window achieving a hemoglobin increase of ≥1.0 g/dL. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by analysis cutoff were censored. The duration of response for participants achieving a hemoglobin increase ≥1.0 g/dL is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 weeks)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Low Dose Group: 0.2 to 0.4 mg/kg | Luspatercept High Dose Group: 0.6 to 1.25 mg/kg
Number analyzed (Participants) | 1 | 13
Days | 126.0 (NA) — NA=standard deviation cannot be calculated for 1 participant. | 118.0 (11.34)

18. Secondary Outcome: Duration of Erythroid Response for Transfusion Dependent (TD) Participants Who Achieved a Transfusion Burden Reduction of ≥50% During a Rolling 12-week Interval
Description: Duration of erythroid response was defined as the time from the first rolling 12-week window achieving a red blood cell (RBC) transfusion burden reduction of ≥50% compared to pretreatment to the last consecutive rolling 12-week window achieving a RBC transfusion burden reduction of ≥50% compared to pretreatment. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by analysis cutoff were censored. The duration of response for participants achieving a RBC transfusion burden reduction of ≥50% compared to pretreatment is presented.
Time Frame: Any 12-week interval during the study (up to approximately 20 weeks)
Population: All participants who received ≥1 dose of study treatment and received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug) and had data available for the analyses. As defined in the clinical study report, the participants with response were pooled into low and high dose groups to reduce the variation of the analyses.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept Low Dose Group: 0.2 to 0.4 mg/kg | Luspatercept High Dose Group: 0.6 to 1.25 mg/kg
Number analyzed (Participants) | 0 | 17
Days |  | 105.0 (17.23)

19. Secondary Outcome: Percent Change From Baseline to End of Treatment in Mean Bone-specific Alkaline Phosphatase (BSAP)
Description: Blood samples were collected at pre-specified time intervals to determine BSAP. The percent change from baseline in BSAP was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for BSAP analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 2 | 3 | 4 | 6 | 6 | 3 | 27
Percent change | 42.6 (14.5) | 3.4 (53) | 8.4 (31.3) | 23.6 (33.3) | 12.7 (53.3) | -20.9 (31.9) | 22.2 (57.7)

20. Secondary Outcome: Percent Change From Baseline to End of Treatment in Mean C-telopeptide of Type I Collagen (CTX)
Description: Blood samples were collected at pre-specified time intervals to determine CTX. The percent change from baseline in CTX was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for CTX analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 6 | 3 | 27
Percent change | -35.1 (10.9) | 15.5 (56.2) | 17.7 (9.3) | 20.1 (20.8) | 0.7 (10.2) | -0.2 (17.2) | 22 (38.1)

21. Secondary Outcome: Percent Change From Baseline to End of Treatment in Serum Iron
Description: Blood samples were collected at pre-specified time intervals to determine serum iron. The percent change from baseline in serum iron was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for serum iron analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 29
Percent change | -15.8 (26.9) | -9.0 (38.0) | 7.8 (15.1) | -12.9 (31.5) | -5.4 (35.8) | -12.4 (18.4) | 2.1 (38.2)

22. Secondary Outcome: Percent Change From Baseline to End of Treatment in Total Iron Binding Capacity (TIBC)
Description: Blood samples were collected at pre-specified time intervals to determine TIBC. The percent change from baseline in TIBC was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for TIBC analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 29
Percent change | 2.9 (7.0) | -1.5 (7.4) | 3.5 (7.8) | -4.9 (11.7) | -2.1 (6.2) | -0.8 (4.3) | 1.3 (12.1)

23. Secondary Outcome: Percent Change From Baseline to End of Treatment in Transferrin
Description: Blood samples were collected at pre-specified time intervals to determine transferrin. The percent change from baseline in transferrin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for transferrin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 29
Percent change | 4.0 (6.7) | -1.5 (6.0) | 3.0 (8.5) | -4.7 (11.3) | -1.0 (7.5) | -1.6 (5.6) | 1.0 (11.5)

24. Secondary Outcome: Percent Change From Baseline to End of Treatment in Soluble Transferrin Receptor
Description: Blood samples were collected at pre-specified time intervals to determine soluble transferrin receptor. The percent change from baseline in soluble transferrin receptor was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for soluble transferrin receptor analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6 | 4 | 29
Percent change | 3.6 (10.9) | -5.9 (5.2) | 10.6 (34.5) | 36.3 (41.3) | 68.2 (60.4) | 83.3 (90.4) | 49.2 (56.9)

25. Secondary Outcome: Percent Change From Baseline to End of Treatment in Ferritin
Description: Blood samples were collected at pre-specified time intervals to determine ferritin. The percent change from baseline in ferritin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for ferritin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 29
Percent change | -18.5 (17.8) | 8.4 (27.2) | -4.5 (14.9) | -23.7 (27.8) | -23.2 (19.4) | -25.2 (22.7) | -23.7 (24.7)

26. Secondary Outcome: Percent Change From Baseline to Day 113 in Serum Non-transferrin Bound Iron (NTBI)
Description: Blood samples were to be collected at pre-specified time intervals to determine NTBI. Baseline was pre-specified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and Day 113
Population: No data were collected for Percent Change From Baseline to Day 113 in Serum NTBI.
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Percent Change From Baseline to Day 113 in Calculated Transferrin Saturation
Description: The calculated transferrin saturation is the ratio of the serum iron concentration and the total iron binding capacity (TIBC) expressed as a percentage. Blood samples were to be collected at pre-specified time intervals for serum iron and TIBC to determine the calculated transferrin saturation. Baseline was pre-specified to be the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and Day 113
Population: No data were collected for Percent Change From Baseline to Day 113 in Calculated Transferrin Saturation.
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hepcidin
Description: Blood samples were collected at pre-specified time intervals to determine hepcidin. The percent change from baseline in hepcidin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for hepcidin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Expansion Cohort: Participants received an initial dose of luspatercept 0.8 mg/kg as an SC injection on Day 1 of the Cycle 1 (Cycle length = 21 days). For each subsequent cycle (up to 5 cycles), the dose was titrated up to a maximum dose of 1.25 mg/kg based on the safety review team (SRT) recommendations.
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 4 | 1 | 10
Percent change | 7.5 (41.1) | 58.4 (141.0) | -4.8 (27.8) | 0.7 (83.3) | -41.2 (12.7) | -13.6 (NA) — Standard deviation could not be calculated for 1 participant | -22.0 (20.9)

29. Secondary Outcome: Percent Change From Baseline to End of Treatment in Reticulocytes
Description: Blood samples were collected at pre-specified time intervals to determine reticulocytes. The percent change from baseline in reticulocytes was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for reticulocyte analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 3 | 6 | 6 | 5 | 6 | 4 | 28
Percent change | -12.41 (19.386) | -2.03 (26.173) | -9.91 (54.978) | 73.38 (61.328) | 25.35 (95.741) | 136.03 (112.261) | 151.26 (435.508)

30. Secondary Outcome: Percent Change From Baseline to End of Treatment in Erythropoietin
Description: Blood samples were collected at pre-specified time intervals to determine erythropoietin. The percent change from baseline in erythropoietin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for erythropoietin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 27
Percent change | -11.18 (55.236) | 10.44 (42.542) | 88.57 (235.111) | 210.69 (311.768) | 97.54 (141.980) | 183.79 (189.662) | 116.25 (245.118)

31. Secondary Outcome: Percent Change From Baseline to End of Treatment in Nucleated Red Blood Cell (nRBC) Count
Description: Blood samples were collected at pre-specified time intervals to determine nRBC count. The percent change from baseline in nRBC count was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for nRBC count analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 2 | 2 | 10
Percent change | -70.19 (42.019) | 17.20 (79.244) | 211.82 (158.143) | 163.63 (178.379) | 176.62 (209.327) | 385.71 (121.218) | 1062.20 (1890.881)

32. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hemoglobin A (Hb A)
Description: Blood samples were collected at pre-specified time intervals to determine Hb A. The percent change from baseline in Hb A was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for Hb A analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6 | 4 | 27
Percent change | -1.96 (7.207) | 308.31 (621.150) | -5.41 (28.623) | -5.00 (16.058) | -22.70 (35.000) | -32.91 (45.256) | -8.46 (20.110)

33. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hemoglobin A2 (Hb A2)
Description: Blood samples were collected at pre-specified time intervals to determine Hb A2. The percent change from baseline in Hb A2 was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for Hb A2 analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 4 | 27
Percent change | 1.14 (21.859) | -14.97 (50.202) | 6.72 (28.515) | -11.49 (50.714) | 26.34 (33.776) | 38.04 (52.758) | 6.15 (18.011)

34. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hemoglobin C (Hb C)
Description: Blood samples were collected at pre-specified time intervals to determine Hb C. The percent change from baseline in Hb C was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for Hb C analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 4 | 27
Percent change | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

35. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hemoglobin D (Hb D)
Description: Blood samples were collected at pre-specified time intervals to determine Hb D. The percent change from baseline in Hb D was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for Hb D analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 4 | 27
Percent change | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

36. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hemoglobin F (Hb F)
Description: Blood samples were collected at pre-specified time intervals to determine Hb F. The percent change from baseline in Hb F was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for Hb F analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 5 | 3 | 27
Percent change | 14.45 (7.734) | -1.96 (13.245) | 37.52 (98.772) | 20.94 (40.153) | 70.89 (57.386) | 308.66 (295.486) | 77.85 (91.560)

37. Secondary Outcome: Percent Change From Baseline to End of Treatment in Hemoglobin S (Hb S)
Description: Blood samples were collected at pre-specified time intervals to determine Hb S. The percent change from baseline in Hb S was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for Hb S analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 4 | 27
Percent change | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)

38. Secondary Outcome: Percent Change From Baseline to End of Treatment in Alpha Globin Gene
Description: Blood samples were collected at pre-specified time intervals to determine alpha globin gene. The percent change from baseline in alpha globin gene was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for alpha globin gene analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 22
Percent change | 42.27 (47.176) | -49.73 (27.324) | -7.11 (79.335) | 389.87 (865.827) | 396.72 (329.535) | -10.85 (54.653) | 1124.14 (2032.635)

39. Secondary Outcome: Percent Change From Baseline to End of Treatment in Beta Globin Gene
Description: Blood samples were collected at pre-specified time intervals to determine beta globin gene. The percent change from baseline in beta globin gene was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for beta globin gene analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 6 | 4 | 21
Percent change | 36.29 (41.033) | -49.17 (29.282) | -15.50 (48.554) | 51.75 (85.913) | 276.26 (215.713) | -6.51 (109.753) | 1056.22 (2400.719)

40. Secondary Outcome: Percent Change From Baseline to End of Treatment in Gamma Globin Gene
Description: Blood samples were collected at pre-specified time intervals to determine gamma globin gene. The percent change from baseline in gamma globin gene was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for gamma globin gene analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 22
Percent change | 81.70 (97.100) | -44.57 (54.656) | -3.32 (109.612) | 468.05 (967.579) | 229.46 (118.097) | -45.40 (32.267) | 1054.42 (1869.511)

41. Secondary Outcome: Percent Change From Baseline to End of Treatment in Haptoglobin
Description: Blood samples were collected at pre-specified time intervals to determine haptoglobin. The percent change from baseline in haptoglobin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for haptoglobin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 5 | 4 | 6 | 4 | 4 | 4 | 13
Percent change | 21.8 (147.4) | 281.0 (434.8) | -16.2 (51.8) | -31.2 (24.9) | 30.3 (181.8) | -55.1 (28.8) | -32.3 (44.3)

42. Secondary Outcome: Percent Change From Baseline to End of Treatment in Indirect Bilirubin
Description: Blood samples were collected at pre-specified time intervals to determine indirect bilirubin. The percent change from baseline in indirect bilirubin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for indirect bilirubin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 29
Percent change | 13.9 (23.7) | -25.2 (18.3) | 4.8 (8.7) | 6.3 (20.3) | 3.7 (21.4) | 2.8 (53.6) | 18.3 (38.7)

43. Secondary Outcome: Percent Change From Baseline to End of Treatment in Lactate Dehydrogenase (LDH)
Description: Blood samples were collected at pre-specified time intervals to determine LDH. The percent change from baseline in LDH was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All participants who received ≥1 dose of study treatment and had data available for LDH analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 4 | 28
Percent change | 0.4 (17.5) | -0.9 (10.5) | 8.7 (25.1) | 29.2 (25.2) | 37.4 (64.5) | 53.8 (68.2) | 45.0 (68.5)

44. Secondary Outcome: Change From Baseline to End of Treatment in Liver Iron Concentration (LIC) For Non-transfusion Dependent (NTD) Participants With Baseline LIC <3 mg/g Dry Weight
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for NTD participants with baseline LIC <3 mg/g dry weight was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The change from baseline to Day 113 in mean LIC for NTD participants with baseline LIC <3 mg/g dry weight is presented.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All NTD participants with baseline LIC <3 mg/g dry weight, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 2 | 1 | 1 | 0 | 0 | 0 | 7
mg/g dry weight | -0.1 (0.09) | -0.5 (NA) — Standard deviation could not be calculated for 1 participant | 0.9 (NA) — Standard deviation could not be calculated for 1 participant |  |  |  | 0.4 (0.67)

45. Secondary Outcome: Change From Baseline to End of Treatment in Liver Iron Concentration (LIC) For Non-transfusion Dependent (NTD) Participants With Baseline LIC ≥3 mg/g Dry Weight
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for NTD participants with baseline LIC ≥3 mg/g dry weight was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The change from baseline to Day 113 in mean LIC for NTD participants with baseline LIC ≥3 mg/g dry weight is presented.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All NTD participants with baseline LIC ≥3 mg/g dry weight, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 4 | 5 | 4 | 2 | 2 | 0 | 3
mg/g dry weight | 0.0 (0.79) | -0.6 (1.22) | -0.6 (2.35) | -1.1 (0.90) | -4.5 (0.18) |  | 0.7 (0.75)

46. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With Baseline Liver Iron Concentration (LIC) of ≥3 mg/g Dry Weight Who Have Demonstrated an LIC Response at End of Treatment
Description: LIC response was defined as a demonstrated LIC reduction of ≥1 mg/g dry weight. Blood samples were collected at pre-specified time intervals to determine LIC in NTD participants with a baseline LIC of ≥3 mg/g dry weight. LIC was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of NTD participants with baseline LIC ≥3 mg/g dry weight who have demonstrated an LIC response is presented.
Time Frame: End of Treatment (up to Day 113)
Population: as for outcome 45
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 4 | 5 | 4 | 2 | 2 | 0 | 3
Percentage of participants | 25.0 [0.6 to 80.6] | 60.0 [14.7 to 94.7] | 50.0 [6.8 to 93.2] | 50.0 [1.3 to 98.7] | 100 [15.8 to 100] |  | 0.0 [0.0 to 70.8]

47. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With Baseline Liver Iron Concentration (LIC) of ≥3 mg/g Dry Weight, Who Have Used Iron Chelation Therapy (ICT), and Who Have Demonstrated an LIC Response at End of Treatment
Description: LIC response was defined as a demonstrated LIC reduction of ≥1 mg/g dry weight. Blood samples were collected at pre-specified time intervals to determine LIC in NTD participants with a baseline LIC of ≥3 mg/g dry weight and who have used ICT. LIC was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of NTD participants with baseline LIC ≥3 mg/g dry weight, who have used ICT, and who have demonstrated an LIC response is presented.
Time Frame: End of Treatment (up to Day 113)
Population: All NTD participants with baseline LIC ≥3 mg/g dry weight, who have used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 2 | 1 | 1 | 0 | 2 | 0 | 2
Percentage of participants | 0.0 [0.0 to 84.2] | 100 [2.5 to 100] | 100 [2.5 to 100] |  | 100 [15.8 to 100] |  | 0.0 [0.0 to 84.2]

48. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With Baseline Liver Iron Concentration (LIC) of ≥3 mg/g Dry Weight, Who Have Not Used Iron Chelation Therapy (ICT), and Who Have Demonstrated an LIC Response at End of Treatment
Description: LIC response was defined as a demonstrated LIC reduction of ≥1 mg/g dry weight. Blood samples were collected at pre-specified time intervals to determine LIC in NTD participants with a baseline LIC of ≥3 mg/g dry weight and who have not used ICT. LIC was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of NTD participants with baseline LIC ≥3 mg/g dry weight, who have not used ICT, and who have demonstrated an LIC response is presented.
Time Frame: End of Treatment (up to Day 113)
Population: All NTD participants with baseline LIC ≥3 mg/g dry weight, who have not used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 2 | 4 | 3 | 2 | 0 | 0 | 1
Percentage of participants | 50.0 [1.3 to 98.7] | 50.0 [6.8 to 93.2] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] |  |  | 0.0 [0.0 to 97.5]

49. Secondary Outcome: Change From Baseline to End of Treatment in Liver Iron Concentration (LIC) For Transfusion Dependent (TD) Participants With Baseline LIC <3 mg/g Dry Weight
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for TD participants with baseline LIC <3 mg/g dry weight was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The change from baseline to Day 113 in mean LIC for TD participants with baseline LIC <3 mg/g dry weight is presented.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All TD participants with baseline LIC <3 mg/g dry weight, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 2 | 9
mg/g dry weight |  |  |  |  | -0.4 (0.21) | 0.2 (0.76) | 0.2 (0.29)

50. Secondary Outcome: Change From Baseline to End of Treatment in Liver Iron Concentration (LIC) For Transfusion Dependent (TD) Participants With Baseline LIC ≥3 mg/g Dry Weight
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for TD participants with baseline LIC ≥3 mg/g dry weight was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The change from baseline to Day 113 in mean LIC for TD participants with baseline LIC ≥3 mg/g dry weight is presented.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 113)
Population: All TD participants with baseline LIC ≥3 mg/g dry weight, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 2 | 1 | 6
mg/g dry weight |  |  | -2.1 (NA) — Standard deviation could not be calculated for 1 participant | -0.7 (1.18) | -0.2 (6.31) | -0.6 (NA) — Standard deviation could not be calculated for 1 participant | -0.6 (1.77)

51. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With Baseline Liver Iron Concentration (LIC) of ≥3 mg/g Dry Weight Who Have Demonstrated an LIC Response at End of Treatment
Description: LIC response was defined as a demonstrated LIC reduction of ≥1 mg/g dry weight. Blood samples were collected at pre-specified time intervals to determine LIC in TD participants with a baseline LIC of ≥3 mg/g dry weight. LIC was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of TD participants with baseline LIC ≥3 mg/g dry weight who have demonstrated an LIC response is presented.
Time Frame: End of Treatment (up to Day 113)
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 2 | 1 | 6
Percentage of participants |  |  | 100 [2.5 to 100] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 33.3 [4.3 to 77.7]

52. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With Baseline Liver Iron Concentration (LIC) of ≥3 mg/g Dry Weight, Who Have Used Iron Chelation Therapy (ICT), and Who Have Demonstrated an LIC Response at End of Treatment
Description: LIC response was defined as a demonstrated LIC reduction of ≥1 mg/g dry weight. Blood samples were collected at pre-specified time intervals to determine LIC in TD participants with a baseline LIC of ≥3 mg/g dry weight and who have used ICT. LIC was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of TD participants with baseline LIC ≥3 mg/g dry weight, who have used ICT, and who have demonstrated an LIC response is presented.
Time Frame: End of Treatment (up to Day 113)
Population: All TD participants with baseline LIC ≥3 mg/g dry weight, who have used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 1 | 3 | 2 | 1 | 5
Percentage of participants |  |  | 100 [2.5 to 100] | 33.3 [0.8 to 90.6] | 50.0 [1.3 to 98.7] | 0.0 [0.0 to 97.5] | 40.0 [5.3 to 85.3]

53. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With Baseline Liver Iron Concentration (LIC) of ≥3 mg/g Dry Weight, Who Have Not Used Iron Chelation Therapy (ICT), and Who Have Demonstrated an LIC Response at End of Treatment
Description: LIC response was defined as a demonstrated LIC reduction of ≥1 mg/g dry weight. Blood samples were collected at pre-specified time intervals to determine LIC in TD participants with a baseline LIC of ≥3 mg/g dry weight and who have not used ICT. LIC was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of TD participants with baseline LIC ≥3 mg/g dry weight, who have not used ICT, and who have demonstrated an LIC response is presented.
Time Frame: End of Treatment (up to Day 113)
Population: All TD participants with baseline LIC ≥3 mg/g dry weight, who have not used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Percentage of participants |  |  |  |  |  |  | 0.0 [0.0 to 97.5]

54. Secondary Outcome: Maximum Concentration (Cmax) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of Cmax. Cmax was defined as the maximum concentration of luspatercept observed after administration. Cmax was based on non-compartmental analysis.
Time Frame: Cycle 1 (21-day cycle): Days 1, 8, 11, and 15; Cycle 2 (21-day cycle): Day 1
Population: The analysis population consisted of all participants who received ≥1 dose of luspatercept and who had available data for the analysis of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
µg/mL | 0.84 (19.95) | 1.52 (21.90) | 2.47 (9.51) | 4.04 (27.45) | 5.73 (29.85) | 6.85 (21.39) | 4.78 (23.60)

55. Secondary Outcome: Time to Maximum Concentration (Tmax) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of Tmax. Tmax was defined as the time to maximum concentration of luspatercept observed after administration. Tmax was based on non-compartmental analysis.
Time Frame: Cycle 1 (21-day cycle): Days 1, 8, 11, and 15; Cycle 2 (21-day cycle): Day 1
Population: The analysis population consisted of all participants who received ≥1 dose of luspatercept and who had available data for the analysis of Tmax.
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
Days | 7.00 [7.00 to 10.00] | 7.00 [7.00 to 9.00] | 7.50 [6.00 to 10.00] | 7.00 [6.00 to 10.00] | 7.00 [6.00 to 7.00] | 7.00 [6.00 to 8.00] | 7.00 [6.00 to 10.00]

56. Secondary Outcome: Area Under the Concentration Time Curve of Luspatercept From Time Zero to Day 21 (AUC0-21)
Description: Blood samples were collected at specified intervals for the determination of AUC0-21. AUC0-21 was defined as the area under the concentration time curve of luspatercept from time zero to Day 21. AUC0-21 was based on non-compartmental analysis and calculated by the linear trapezoidal method.
Time Frame: Cycle 1: Days 1, 8, 11, and 15; Day 22 (Cycle 2 Day 1). Cycles 1 and 2 are 21-day cycles
Population: The analysis population consisted of all participants who received ≥1 dose of luspatercept and who had available data for the analysis of AUC0-21.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day●µg/mL
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 29
day●µg/mL | 11.68 (20.53) | 20.66 (22.79) | 31.43 (12.16) | 54.30 (26.66) | 70.39 (34.84) | 93.79 (23.75) | 62.70 (29.58)

57. Secondary Outcome: Terminal Elimination Half Life (t½) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of t½. t½ was defined as the time required to divide the serum concentration of luspatercept by two after reaching pseudo-equilibrium. t½ was based on non-compartmental analysis.
Time Frame: Cycle 1 (21-day cycle): Days 1, 8, 11, and 15; Cycle 2 (21-day cycle): Days 1 and 8; Cycles 4 and 5 (21-day cycles): Days 1, 8, and 15; study follow-up on Days 113, 141, and 169
Population: The analysis population consisted of all participants who received ≥1 dose of luspatercept and who had available data for the analysis of t½.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 6 | 4 | 25
Days | 11.56 (27.52) | 10.12 (34.41) | 9.65 (21.48) | 11.22 (19.94) | 9.42 (25.73) | 10.37 (13.34) | 10.79 (24.19)

58. Secondary Outcome: Apparent Terminal Rate Constant (Lambda z) of Luspatercept
Description: Blood samples were collected at specified intervals for the determination of apparent terminal rate constant. Apparent terminal rate constant was defined as the amount of luspatercept that was eliminated from the body during a given period of time and was calculated by linear regression of the terminal portion of the log-concentration-time curve in serum. Apparent terminal rate constant was based on non-compartmental analysis.
Time Frame: as for outcome 57
Population: The analysis population consisted of all participants who received ≥1 dose of luspatercept and who had available data for the analysis of apparent terminal rate constant.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/Day
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
Number analyzed (Participants) | 6 | 6 | 6 | 4 | 6 | 4 | 25
1/Day | 0.06 (27.52) | 0.07 (34.41) | 0.07 (21.48) | 0.06 (19.94) | 0.07 (25.73) | 0.07 (13.34) | 0.06 (24.19)

ADVERSE EVENTS:
Time Frame: Up to approximately 20 weeks
Description: All-cause mortality was reported on all allocated participants. Serious and non-serious adverse events were reported on all participants who received ≥1 dose of study treatment.
Arm/Group | Luspatercept 0.2 mg/kg | Luspatercept 0.4 mg/kg | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg | Expansion Cohort
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/29
Other Adverse Events (participants affected / at risk) | 5/6 | 6/6 | 5/6 | 6/6 | 6/6 | 5/5 | 25/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.2 mg/kg (N=6) | Luspatercept 0.4 mg/kg (N=6) | Luspatercept 0.6 mg/kg (N=6) | Luspatercept 0.8 mg/kg (N=6) | Luspatercept 1.0 mg/kg (N=6) | Luspatercept 1.25 mg/kg (N=5) | Expansion Cohort (N=29)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.2 mg/kg (N=6) | Luspatercept 0.4 mg/kg (N=6) | Luspatercept 0.6 mg/kg (N=6) | Luspatercept 0.8 mg/kg (N=6) | Luspatercept 1.0 mg/kg (N=6) | Luspatercept 1.25 mg/kg (N=5) | Expansion Cohort (N=29)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythroblastosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 2 (2) | 2 (3) | 11 (28)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Peripheral swelling (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 2 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (8)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parvovirus B19 infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood 25-hydroxycholecalciferol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (16) | 0 (0) | 2 (3) | 7 (16)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (7) | 4 (31) | 2 (7) | 3 (4) | 14 (44)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 7 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 2 (2) | 3 (8) | 0 (0) | 2 (2) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (7) | 0 (0) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (7) | 3 (8) | 4 (8) | 2 (3) | 8 (21)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (3) | 1 (4) | 1 (1) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or disclosure of study results will be permitted except as specified in a separate, written, agreement between the sponsor and the investigator(s).

DOCUMENTS (2):
  • Study Protocol (2014-11-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT01749540/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT01749540/SAP_001.pdf